CLINICAL TRIAL: NCT07097389
Title: In Vivo Human Study on Commercial Cellobiose as a Potential Prebiotic Candidate
Acronym: C-prebiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manxi Huang (Other)
Responsible Party: Sponsor-Investigator, Manxi Huang, PhD Candidate, Department of Food and Nutritional Sciences, University of Reading
Organization: University of Reading (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UREC24/20
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Gut -Microbiota; As a Preliminary Study, Healthy Population's Gut Microbiota is Studied to See if Cellobiose Supplementation is Altering the Microbial Community or Not
Keywords: cellobiose; preliminary in vivo human study
MeSH Terms: interventions — Cellobiose; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Maltodextrin (Placebo Comparator): Participants receive 5 g/day for the first 7 days and 10 g/day maltodextrin for the rest of the 21 days as a non-prebiotic control.
  Interventions: Dietary Supplement: Maltodextrin (Placebo)
- Orafti P95 (oligofructose P95) (Active Comparator): Healthy adult volunteers will consume 5 g/day of Orafti P95 (oligofructose, Beneo GmbH) mixed in water for the first 7 days, and consume 10 g/day of Orafti P95 (oligofructose, Beneo GmbH) mixed in water for the rest of the 21 days.
  Interventions: Dietary Supplement: Oligofructose P95
- Cellobiose (Experimental): Participants receive 5g/day for the first 7 days and 10 g/day cellobiose for 21 days.
  Interventions: Dietary Supplement: Cellobiose

INTERVENTIONS:
Dietary Supplement: Cellobiose — Cellobiose powder (Savanna Ingredients GmbH), 5 g per day and 10 g per day, mixed into ~200 mL water and taken orally with breakfast for the first 7 days and the rest of the 21 days.
  Arms: Cellobiose
Dietary Supplement: Oligofructose P95 — Oligofructose (Orafti® P95, Beneo GmbH), 5 g per day and 10 g per day, dissolved in ~200 mL water and taken orally with breakfast for the first 7 days and the rest of the 21 days.
  Arms: Orafti P95 (oligofructose P95)
Dietary Supplement: Maltodextrin (Placebo) — Maltodextrin powder (Special Ingredients Limited), 5 g per day and 10 g per day, dissolved in ~200 mL water and taken orally with breakfast for the first 7 days and the rest of the 21 days.
  Arms: Maltodextrin

SUMMARY:
The goal of this project is to investigate whether cellobiose, a type of sugar, has a beneficial effect on gut health when consumed by humans. Cellobiose will be obtained from spent coffee grounds through enzymatic modification, repurposing waste biomass for a potentially valuable purpose. The study will only focus on conducting in vivo human trials using a commercial form of cellobiose from Savanna Ingredients GmbH, which has recently been approved as a novel food by the EU (https://eur-lex.europa.eu/eli/reg_impl/2023/943/oj)

We will also be testing two other commercial products: Orafti® P95, an oligofructose-based product from Beneo GmbH, and maltodextrin from Special Ingredients Limited. These products will be compared to evaluate their potential in promoting gut health by nourishing beneficial bacteria, The study will involve feeding these products to volunteers and observing their impact on gut health.

The key questions this project aims to address include:

* Does cellobiose, exhibit any gut health promoting effects in humans?
* How does cellobiose compare to other commercial prebiotic products, such as Orafti® P95, in terms of its effects on gut health?

To conduct the study, volunteers will be provided with the three different products to consume over a specified period. Their faecal samples will be collected at various points to assess changes in gut microbiota composition and other indicators of gut health. This will involve close monitoring of participants' health and adherence to ethical guidelines to ensure their safety and well-being throughout the study.

Overall, this project seeks to expand our understanding of the potential health benefits of cellobiose and other prebiotic carbohydrates. It aims to provide valuable insights into the role of these substances in promoting gut health.

DETAILED DESCRIPTION:
In this randomised, double-blinded, parallel-group trial, the investigators will enroll 36 healthy adult volunteers and randomise them 1:1:1 to one of three dietary-supplement arms. Participants will consume their assigned product once daily-5 g during a one-week adaptation phase followed by 10 g/day for a three-week intervention phase. Faecal samples will be collected at baseline (Visit 1) and at study completion (Visit 5). Total bacterial counts will be determined by fluorescence in situ hybridisation coupled with flow cytometry (FISH-FLOW), and short-chain fatty acid concentrations quantified by gas chromatography-flame ionisation detection (GC-FID).

The primary outcomes are the change from baseline to Visit 5 in (1) absolute abundance of Bifidobacterium spp. and Lactobacillus spp., and (2) total faecal short-chain fatty acid concentration. Secondary outcomes include gut microbiota diversity metrics (α- and β-diversity) and daily gastrointestinal symptom incidence. Exploratory outcomes will assess correlations between shifts in specific bacterial taxa and metabolite profiles, as well as changes in the abundance of other key genera.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

1. Participants aged 18 years old and above
2. Participants are willing to comply with the study instructions
3. Participants have a stool frequency of at least 3 bowel movements per week
4. Participants are healthy at the time of signing the consent form

Exclusion criteria:

1. Not pregnant or planning to be pregnant
2. Previously or currently diagnosed gastrointestinal diseases and disorders that might affect the gut environment.
3. Food allergies or intolerances
4. Previously or currently diagnosed with cancer or taking a long-term medication.
5. Use of medication (e.g, antibiotics, aspirin, proton pump inhibitors) influencing gastrointestinal function (8 weeks before intervention)
6. Participants are currently involved or will be involved in another clinical or food study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change in absolute abundance of faecal Bifidobacterium spp. and Lactobacillus spp. | Baseline (Day 0; Visit 1) to end of the intervention period (Day 28; Visit 5)
  Absolute abundance of Bifidobacterium spp. and Lactobacillus spp. in faecal microbiota, determined by 16S rRNA gene sequencing (Illumina NGS sequencing) and FLOW-FISH for total bacterial counts
Change in total faecal short-chain fatty acid concentration | Baseline (Day 0; Visit 1) to end of the intervention(Day 28; Visit 5)
  Sum of acetate, propionate, and butyrate concentrations in faecal samples, measured by GC-MS.

SECONDARY OUTCOMES:
Magnitude and pattern of overall gut-microbiota shifts from V1 to V5 | Baseline (V1) through end-point (V5) of the 28-day intervention
  The magnitude and pattern of gut-microbiota compositional shifts from baseline (V1) to end-point (V5), quantified by each subject's within-pair Bray-Curtis distance and visualized via PCoA, with statistical significance assessed by a paired PERMANOVA (Visit as fixed effect, Subject as blocking factor).
Number of participants with Gastrointestinal Tolerability & Safety | Days 1 through 28 of the intervention period
  Participants completed a daily diary during Days 1-28 of the intervention in which they:
  Recorded the time of product ingestion.
  Tick-boxed any GI symptoms each day from the following list:
  Bloating, Gas/Flatulence, Abdominal pain/cramps, Diarrhoea
  Nausea, Vomiting, Frequency of bowel movements, Constipation, Changes in stool consistency
  If "Changes in stool consistency" was ticked, they described the change in a free-text field (e.g., "looser," "harder").

OTHER OUTCOMES:
SCFA-Microbe Correlations & Other Genus Fold-Changes | Baseline (V1) through end-point (V5) of the 28-day intervention.
  SCFA-Microbe Correlations
  For each subject, compute log₂-fold-changes (V5 vs V1) in stool acetate, propionate, and butyrate.
  Compute Spearman correlation coefficients (ρ) and 95 % CIs between each SCFA change and log₂-fold-changes in Bifidobacterium and Lactobacillus.
  Fold-Changes in Other Key Genera
  Calculate mean log₂-fold-changes ± 95 % CIs (V5 vs V1) for the following genera: Faecalibacterium, Blautia, Roseburia, Bacteroides,
  No formal hypothesis tests-these are reported as effect-size estimates only.

CONTACTS AND LOCATIONS:
Overall Officials: Bob Rastall, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the primary and secondary outcomes (microbiome absolute counts, SCFA concentrations, GI symptom diaries), along with the study protocol and statistical analysis plan, will be made available to qualified researchers beginning six months after publication. Requests can be submitted to the corresponding author (r.a.rastall@reading.ac.uk) and will require a signed data-use agreement. Data will be shared in CSV format.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Six months after publication, with data available for up to five years thereafter.
Access Criteria: The data will be available to qualified researchers who submit a reasonable research proposal and execute a data-use agreement.